CLINICAL TRIAL: NCT01059539
Title: A Long-term Open-label Study of the Safety and Tolerability of Cariprazine in Patients With Bipolar I Disorder
Brief Title: Long-term Safety and Tolerability of Cariprazine for Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Gedeon Richter Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RGH-MD-36
Record Dates: First submitted 2010-01-27; First posted 2010-02-01 (Estimated); Results first posted 2019-06-13 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-05

CONDITIONS: Bipolar I Disorder
Keywords: Mania; Acute mania; Bipolar I disorder
MeSH Terms: conditions — Mania | interventions — cariprazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cariprazine 3-12 mg/day for 16 weeks (Experimental): Participants received cariprazine 1.5 mg orally on Day 1 and cariprazine 3.0 mg orally on Days 2 and 3. Starting on Day 4, the dose could be increased in increments of 3 mg every 2 days up to a maximum dose of 12 mg, if the response was not adequate and there were no tolerability issues based on the judgment of the principal investigator.
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine — Cariprazine was supplied in capsules.
  Other Names: RGH-188

SUMMARY:
The objective of this study is to evaluate the long-term safety, tolerability, and pharmacokinetics of cariprazine in patients with bipolar I disorder.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have provided informed consent prior to any study specific procedures.
* Patients currently meeting the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR) criteria for bipolar I disorder as confirmed by the Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (SCID).
* Patients who experienced a manic or mixed episode that required treatment within the past 12 months.
* Patients with normal physical examination, laboratory, vital signs, and electrocardiogram (ECG).

Exclusion Criteria:

* Patients with a DSM-IV-TR diagnosis of an axis I disorder other than bipolar I disorder.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 403 (Actual)
Dates: Start 2010-02-28 (Actual); Primary Completion 2012-02-29 (Actual); Study Completion 2012-02-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Diaz, MD, Study Director — Forest Laboratories
Locations (35):
- United States (24):
  - Forest Investigative Site 015, Springdale, Arkansas
  - Forest Investigative Site 010, Carson, California
  - Forest Investigative Site 020, Cerritos, California
  - Forest Investigative Site 009, Escondido, California
  - Forest Investigative Site 004, Garden Grove, California
  - Forest Investigative Site 016, San Diego, California
  - Forest Investigative Site 007, Santa Ana, California
  - Forest Investigative Site 023, Washington D.C., District of Columbia
  - Forest Investigative Site 001, Bradenton, Florida
  - Forest Investigative Site 006, Fort Lauderdale, Florida
  - Forest Investigative Site 013, Kissimmee, Florida
  - Forest Investigative Site 021, Rockville, Maryland
  - Forest Investigative Site 024, Flowood, Mississippi
  - Forest Investigative Site 022, Creve Coeur, Missouri
  - Forest Investigative Site 003, Saint Charles, Missouri
  - Forest Investigative Site 025, St Louis, Missouri
  - Forest Investigative Site 012, Las Vegas, Nevada
  - Forest Investigative Site 002, Willingboro, New Jersey
  - Forest Investigative Site 005, Cincinnati, Ohio
  - Forest Investigative Site 011, Oklahoma City, Oklahoma
  - Forest Investigative Site 017, Austin, Texas
  - Forest Investigative Site 014, Austin, Texas
  - Forest Investigative Site 018, DeSoto, Texas
  - Forest Investigative Site 019, Houston, Texas
- Hungary (5):
  - Forest Investigative Site 309, Gyula, Bekes County
  - Forest Investigative Site 301, Budapest
  - Forest Investigative Site 302, Budapest
  - Forest Investigative Site 306, Nyíregyháza
  - Forest Investigative Site 308, Szombathely
- Poland (5):
  - Forest Investigative Site 402, Tuszyn, Kodz
  - Forest Investigative Site 404, Katowice, Silesian
  - Forest Investigative Site 407, Gdansk
  - Forest Investigative Site 408, Gmina Świecie
  - Forest Investigative Site 401, Gorlice
- Forest Investigative Site 505, Barcelona, Spain

REFERENCES:
- [Derived] Ketter TA, Sachs GS, Durgam S, Lu K, Starace A, Laszlovszky I, Nemeth G. The safety and tolerability of cariprazine in patients with manic or mixed episodes associated with bipolar I disorder: A 16-week open-label study. J Affect Disord. 2018 Jan 1;225:350-356. doi: 10.1016/j.jad.2017.08.040. Epub 2017 Aug 18. PMID 28843918

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cariprazine 3-12 mg/Day for 16 Weeks
Started | 403
Completed | 132
Not Completed | 271
Not completed — Adverse Event | 66
Not completed — Insufficient Therapeutic Response | 26
Not completed — Protocol Violation | 55
Not completed — Withdrawal of Consent | 80
Not completed — Lost to Follow-up | 42
Not completed — Reason Not Specified | 2

BASELINE CHARACTERISTICS:
Population: Safety population: All enrolled participants who took at least 1 dose of investigational product.
Arm/Group | Cariprazine 3-12 mg/Day for 16 Weeks
Number analyzed (Participants) | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 230
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32
  Not Hispanic or Latino | 370
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 182
  White | 206
  More than one race | 3
  Unknown or Not Reported | 0
Weight [Mean (Standard Deviation); unit: kg] | 86.52 (17.83)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.21 (5.34)
Waist circumference [Mean (Standard Deviation); unit: cm] | 97.86 (14.05)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the YMRS Total Score at Week 16
Description: The Young Mania Rating Scale (YMRS) is an 11-item scale that assesses manic symptoms based on the patient's perception of his or her condition over the previous 48 hours, as well as the physician's clinical observations during the interview. The 11 items are elevated mood, increased motor activity-energy, sexual interest, sleep, irritability, rate and amount of speech, language-thought disorder, content, disruptive-aggressive behavior, appearance, and insight. The severity of each item is rated on a 5-point (0-4) or a 9-point (0-8) scale. The total score of all 11 items can range from 0 to 60. A higher score indicates worse manic symptoms. A negative change score indicates improvement.
Time Frame: Baseline to Week 16
Population: Intent-to-treat population: All enrolled participants who took at least 1 dose of investigational product and who had a Baseline and at least 1 post-baseline assessment of the Young Mania Rating Scale.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cariprazine 3-12 mg/Day for 16 Weeks
Number analyzed (Participants) | 399
Units on a scale | -15.2 (9.2)

2. Secondary Outcome: Change From Baseline in the MADRS Total Score at Week 16
Description: The Montgomery-Asberg Depression Rating Scale (MADRS) is a clinician-rated scale that evaluates the patient's depressive symptomatology during the previous week. Patients are rated on 10 items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each item is scored on a 7-point (0-6) scale. The total score can range from 0 to 42. A higher score indicates greater depressive symptomatology. A negative change score indicates improvement.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Cariprazine 3-12 mg/Day for 16 Weeks
Number analyzed (Participants) | 399
Units on a scale | -1.6 (7.5)

ADVERSE EVENTS:
Description: Safety population: All enrolled participants who took at least 1 dose of investigational product.
Arm/Group | Cariprazine 3-12 mg/Day for 16 Weeks
All-Cause Mortality (participants affected / at risk) | 0/402
Serious Adverse Events (participants affected / at risk) | 34/402
Other Adverse Events (participants affected / at risk) | 293/402
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine 3-12 mg/Day for 16 Weeks (N=402)
Mania (Psychiatric disorders) | 9
Depression (Psychiatric disorders) | 5
Akathisia (Psychiatric disorders) | 3
Suicidal ideation (Psychiatric disorders) | 2
Suicide attempt (Psychiatric disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Anxiety (Psychiatric disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Bipolar I disorder (Psychiatric disorders) | 1
Bradycardia (Cardiac disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Dermal cyst (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Hypersensitivity (Immune system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Intentional overdose (Injury, poisoning and procedural complications) | 1
Non-cardiac chest pain (Respiratory, thoracic and mediastinal disorders) | 1
Panic attack (Psychiatric disorders) | 1
Paranoia (Psychiatric disorders) | 1
Pneumonia (Infections and infestations) | 1
Social stay hospitalization (Social circumstances) | 1
Tremor (Nervous system disorders) | 1
Large intestinal obstruction/Large bowel obstruction (Gastrointestinal disorders) | 1
Psychotic disorder/Increased psychosis (Psychiatric disorders) | 1
Psychotic disorder/Psychosis (Psychiatric disorders) | 1
Mania/Increased mania (Psychiatric disorders) | 1
Mania/Worsening of mania (Psychiatric disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cariprazine 3-12 mg/Day for 16 Weeks (N=402)
Constipation (Gastrointestinal disorders) | 44
Diarrhoea (Gastrointestinal disorders) | 22
Dyspepsia (Gastrointestinal disorders) | 38
Nausea (Gastrointestinal disorders) | 42
Toothache (Gastrointestinal disorders) | 35
Vomiting (Gastrointestinal disorders) | 25
Weight increased (Investigations) | 25
Back pain (Musculoskeletal and connective tissue disorders) | 32
Akathisia (Nervous system disorders) | 129
Extrapyramidal disorder (Nervous system disorders) | 28
Headache (Nervous system disorders) | 69
Sedation (Nervous system disorders) | 24
Tremor (Nervous system disorders) | 31
Insomnia (Psychiatric disorders) | 27
Restlessness (Psychiatric disorders) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All data generated in this study will be the property of Forest Research Institute, Inc. An integrated clinical and statistical report will be prepared at the completion of the study. Publication of the results by the Investigator will be subject to mutual agreement between the Investigator and Forest Research Institute, Inc.